CLINICAL TRIAL: NCT00233246
Title: Study of Hemostasis and Invasive Procedures (SHIP: A TMH CTN Study)
Brief Title: Fresh-Frozen Plasma Infusions to Reduce Risk of Bleeding Related to Invasive Procedures
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study never activated
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Transfusion Medicine/Hemostasis Clinical Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Prevention
Other Study IDs: 326; U01HL072299 (NIH); U01HL072028 (NIH); U01HL072072 (NIH); U01HL072191 (NIH); U01HL072196 (NIH); U01HL072248 (NIH); U01HL072289 (NIH); U01HL072290 (NIH); U01HL072291 (NIH); U01HL072305 (NIH); U01HL072331 (NIH); U01HL072346 (NIH); U01HL072355 (NIH); U01HL072359 (NIH); U01HL072283 (NIH)
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Blood Coagulation Disorders
MeSH Terms: conditions — Blood Coagulation Disorders

INTERVENTIONS:
Procedure: FFP Infusion

SUMMARY:
This study will compare patients with mild to moderate prolongation of the INR test who receive FFP infusions prior to invasive hepatobiliary procedures for bleeding complications to patients who do not receive FFP infusions. Bleeding complications will be defined as meeting one or more of the following:

1. Intrahepatic hematoma greater than 1 ml/kg of patient weight as seen on post-procedure ultrasound examination performed between 4 to 30 hours after the procedure.
2. Greater than 1.6g/dL hemoglobin decline measured within 4 to 30 hours post-procedure compared with the pre-procedure value, in the absence of another identified bleeding source to account for the hemoglobin drop.
3. Need for transfusion of packed red blood cells for procedure-related bleeding while in the study.

The secondary endpoints of this study will be: 1) The need to perform subsequent procedures (angiography, embolization, additional imaging study including computerized tomography (CT) scan, surgery) to diagnose or to arrest procedure-related bleeding OR the need for subsequent medical therapies (FFP, coagulation factor concentrates, anti-fibrinolytics) to treat procedure-related bleeding between time of procedure and the end of patient's time in the study. If necessary, the relationship of procedure or therapy to procedure-related bleeding will be assessed by an adjudication panel; 2) The predictive value of INR; 3) The effect of study treatment on change in INR; 4) The cost of preventing one bleed; 5) The predictors of bleeding other than INR; 6) The number of transfusion-associated adverse events encountered to prevent one bleed; and 7) The effect of treatment on bleeding grade.

DETAILED DESCRIPTION:
BACKGROUND:

It is important to determine whether or not prophylactic FFP is necessary for patients with mild to moderate elevation of the INR who require an invasive procedure. It is also important to establish whether routine pre-procedure coagulation tests are predictive of bleeding outcomes at the time of a significant invasive procedure. Although prophylactic FFP is often given to such patients before invasive procedures, there is little evidence to show that pre-procedure INR in this range is predictive of procedure-related bleeding or that prophylactic FFP reduces this risk.

DESIGN NARRATIVE:

After obtaining consent and verifying eligibility requirements, the study staff will randomize the patient to one of two treatment groups. One group will receive a prophylactic FFP infusion before the hepatobiliary procedure. The other group will not receive prophylactic FFP.

The dose of FFP will be approximately 10 ml/kg. The dose of FFP for each patient will be determined in one of two ways in accordance with local policies: 1) rounding to the nearest integer number of units (Method 1); or 2) using split units (Method 2). The method chosen may vary between patients (e.g., a physician might decide to dose adult patients by rounding to the nearest integer number of units and to dose pediatric patients using split units).

Method 1: The dose of FFP will be the number of units that comes closest to a dose of 10 ml/kg, determined as follows: nearest integer to (10 x weight in kg)/200. Decimals .5 and higher should be rounded up to the next integer. Decimals less than .5 should be rounded down (e.g., a 70 kg patient would receive 4 units, while a 69 kg patient would receive 3 units).

Method 2: The dose of FFP will be chosen in order to come as close as possible to a dose of 10 ml/kg, and can contain either full units, split units, or a combination thereof.

After the FFP infusion (if any) and within 2 hours prior to the hepatobiliary procedure, blood will be drawn for laboratory tests and for the repository. Although Study of Hemostasis and Invasive Procedures (SHIP) will not be a truly blinded study, the clinicians performing the hepatobiliary procedure and the radiology team performing the post-procedure ultrasound will not be told whether the participant received prophylactic FFP. They will also not know the results of the immediate pre-procedure Prethrombin Time (PT)/INR and Partial Thomboplastin Time (PTT) tests.

Participants in the study may not be treated with any other systemic hemostatic agents prior to the procedure. Local hemostatic treatments may be used during the procedure, according to standard practice. The invasive hepatobiliary procedure techniques, all other concomitant treatments and interventions, and all post-procedure treatments and interventions are at the discretion of the treating physicians. Participants will be followed for clinical evidence of bleeding and will be treated as needed for any bleeding that may occur.

Repository samples will only be used for genetic and protein tests of hemostasis, coagulation, and fibrinolysis.

SHIP is designed as a one-sided non-inferiority study. The null hypothesis is that the proportion of patients not given prophylactic FFP who meet the criteria for the bleeding endpoint is at least .04 higher than the proportion of patients given prophylactic FFP who meet the criteria for the bleeding endpoint. The goal of this study is to determine whether there is strong evidence that the difference between the two treatment plans is not that large.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing one of the following percutaneous abdominal or transjugular invasive procedures: liver biopsy; liver-biliary abscess drainage; biliary tree drainage; or radio-frequency ablation of hepatic tumor
* Platelet count greater than or equal to 70,000/microliter
* INR greater than or equal to 1.3 and less than or equal to 1.9 (must not be based on a sample drawn within 24 hours of any prior FFP treatment)
* A PTT less than or equal to 50 sec

Exclusion Criteria:

* Use of warfarin, heparin, low molecular weight heparin, or other anticoagulant therapy within 5 days of the planned procedure (exceptions: prophylactic heparin injections into central venous catheters for catheter maintenance, prophylactic heparin (standard or low-dose) for prevention of deep venous thrombosis, and/or aspirin)
* History of severe allergic reaction to plasma products
* Use of any of the following second-generation anti-platelet agents: abciximab, tirofiban, clopidogrel, or ticlopidine
* Currently receiving any dialysis
* History of clinically significant bleeding diathesis, including Hemophilia A or B, von Willebrand's Disease, or congenital Factor VII deficiency
* Known history of a coagulation-factor inhibitor within the month prior to the procedure (In the absence of a known history, testing is not required)
* Active major bleeding; bleeding from gastrointestinal, pulmonary, mouth/throat, genito-urinary tract, or central nervous system sites (excludes guaiac positive stool sample without gross blood or melena, minor epistaxis, minor gum bleeding, microscopic hematuria, superficial bruises, normal menses, or minor vaginal spotting)
* Pediatric patients requiring sedation in order to undergo a post-procedure ultrasound examination
* Already received FFP in the 24 hours before the planned invasive procedure

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-03

PRIMARY OUTCOMES:
Clinically significant bleeding (measured 4 to 30 hours after invasive hepatobiliary procedure)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Assmann, PhD, Principal Investigator — New England Research Institutes, Inc.; Mark Brecher, MD, Principal Investigator — University of North Carolina Hospital; George Buchanan, MD, Principal Investigator — University of Texas SW Medical Center; James Bussel, MD, Principal Investigator — Weill Medical College of Cornell University; John Hess, MD, MPH, Principal Investigator — University of Maryland, Baltimore; Christopher D. Hillyer, MD, Principal Investigator — Emory University; Barbara Konkle, MD, Principal Investigator — University of Pennsylvania; David Kuter, MD, Principal Investigator — Massachusetts General Hospital; Jeffrey McCullough, MD, Principal Investigator — University of Minnesota; Janice McFarland, MD, Principal Investigator — Blood Center of SE Wisconsin; Paul Ness, MD, Principal Investigator — Johns Hopkins University; Thomas Ortel, MD, PhD, Principal Investigator — Duke University; Sherrill J. Slichter, MD, Principal Investigator — Puget Sound Blood Center Div of Research; Ronald Strauss, MD, Principal Investigator — University of Iowa; Darrell Triulzi, MD, Principal Investigator — University of Pittsburgh Presbyterian and Shadyside Hospital; James R. Stubbs, MD, Principal Investigator — Mayo Clinic
Locations (15):
- United States (15):
  - Emory University, Atlanta, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Weill Medical College of Cornell University, New York, New York
  - University of North Carolina Hospital, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Presbyterian and Shadyside Hospital, Pittsburgh, Pennsylvania
  - University of Texas SW Medical Center, Dallas, Texas
  - Puget Sound Blood Center Div of Research, Seattle, Washington
  - Blood Center of SE Wisconsin, Milwaukee, Wisconsin